CLINICAL TRIAL: NCT02983084
Title: SmartWire Multiforce Archwire Clinical Trial
Brief Title: Orthodontic Archwire Comparison Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ormco Corporation (Industry)
Collaborators: Indiana University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1608063565
Record Dates: First submitted 2016-11-29; First posted 2016-12-06 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Malocclusion
Keywords: Orthodontic wires; Root resorption
MeSH Terms: conditions — Malocclusion; Root Resorption

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Multiforce (Experimental): Variable modulus version of a current orthodontic archwire
  Interventions: Device: Orthodontic archwire
- CuNiTi A (Active Comparator): .016" current orthodontic archwire
  Interventions: Device: Orthodontic archwire
- CuNiTi B (Active Comparator): 0.014" and 0.018" current orthodontic archwire sequence
  Interventions: Device: Orthodontic archwire

INTERVENTIONS:
Device: Orthodontic archwire — Archwire used to align teeth in an orthodontic fixed appliance
  Other Names: Multiforce CuNiTi; CuNiTi; Copper Nickel Titanium

SUMMARY:
The purpose of this randomized clinical trial (RCT) is to compare traditional CuNiTi archwires and a recently marketed multiforce version of the same material for the initial alignment and leveling of dental arches, as well as the expression of EARR in adult orthodontic patients.

DETAILED DESCRIPTION:
This is a randomized clinical trial utilizing multiforce and CuNiTi orthodontic archwires to align and level dental arches and compare their results. A three group double blind parallel single site study at IUSD will be used.

Patients that meet the inclusion and exclusion criteria will be recruited from the IUSD orthodontic clinic. The subjects will be randomly assigned to one of the three groups by the study statistician. Subjects, examiners providing subject treatment, and examiners measuring study outcomes will be blinded to treatment assignment.

Study population indicates a sample size of 105 subjects, each group containing 35 clinical subjects.

Patients will be treated with Ormco Titanium Orthos fixed appliances and defined archwire sequence according to a clinical protocol. During the six-month study period, subjects will be seen approximately every 4 (four) weeks for regular standard of care appointments that will include archwire monitoring, photography and questionnaire completions. Final study records will be taken at the end of the study period.

ELIGIBILITY:
Inclusion Criteria:

* Adult >14yrs of age
* Amenable to treatment with metal brackets
* Crowding of 3-8mm in one or both arches (non-extraction treatment)
* Overbite >3mm
* Read and speak English without a translator
* Individuals in good general health at the discretion of the investigator(s)

Exclusion Criteria:

* Medical/Dental History (Hx):

  * Documented metabolic disorder(s)
  * Nickel allergy
  * Bisphosphonate treatment
  * Amelogenesis, dentinogenesis or osteogenesis imperfect
  * Active caries or periodontal disease
  * Root resorption (moderate to severe)
  * Patients who are pregnant or breast feeding or plan to be pregnant during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2016-12-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Alignment of dental arches | Initial six months of treatment
  Tooth alignment rate in response to force from archwire measured in mm on dental models

SECONDARY OUTCOMES:
Leveling of dental arches | Initial six months of treatment
  Depth of the Curve of Spee (CoS): percent correction during the six month initial alignment
Expression of external apical root resorption (EARR) | Initial six months of treatment
  Amount of root resorption in response to force from archwire calculated in 3D from the CBCT

CONTACTS AND LOCATIONS:
Overall Officials: Kelton T Stewart, DDS, MS, Principal Investigator — Indiana Unversity
Locations (1):
- IUSD Orthodontic Clinic, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No